CLINICAL TRIAL: NCT00475176
Title: Effects of S-Adenosyl Methionine (SAMe) on Viral and Cell Signaling Response to Combination Therapy for Chronic Hepatitis C
Brief Title: S-Adenosyl Methionine (SAMe) to Treat Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jay Hoofnagle, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070143; 07-DK-0143 (Other: NIHCC); 07-DK-0143 (Other: National Institutes of Health Clinical Center)
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2013-07-05 (Estimated); Last update posted 2013-07-05 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C Virus Genotype 1; Non-Responders; SAMe; Natural Killer Cells; Interferon Signaling; Ribavirin; Peginterferon; Hemolysis; STAT; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hemolysis; Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin; S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-Adenosyl Methionine (Experimental)
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: S-adenosyl methionine for Chronic Liver Disease

INTERVENTIONS:
Drug: Peginterferon alfa-2a
Drug: Ribavirin
Drug: S-adenosyl methionine for Chronic Liver Disease

SUMMARY:
This study will examine the effectiveness of S-adenosyl methionine (SAMe) in combination with peginterferon and ribavirin for treating hepatitis C virus. One out of three patients with hepatitis C develops cirrhosis of the liver, which can lead to liver failure or liver cancer. SAMe is a nutritional supplement that is made naturally in all cells of the body and acts to improve how the body handles stress. In laboratory experiments with liver cells, SAMe decreases the injury caused by liver toxins and improves the ability of interferon to block hepatitis C virus.

Patients 18 years of age and older with hepatitis C infection who did not respond successfully to prior treatment with interferon and ribavirin or peginterferon and ribavirin may be eligible for this study.

Participants receive the following treatment:

* Peginterferon (given by injection) and ribavirin (taken by mouth) for 2 weeks
* Washout period (no medications) for 4 weeks
* SAMe (taken by mouth) for 2 weeks
* Peginterferon, ribavirin and SAMe for 12-48 weeks, depending on patient response to treatment.

Participants have a thorough physical evaluation before beginning treatment and again at the study's end. After starting treatment, patients return for clinic visits and blood tests weekly for the first several weeks, then less frequently (at 2-week, then 4-week and 8-week intervals until up to 72 weeks) to monitor symptoms, drug side effects, hepatitis C virus levels, liver enzyme levels and immune responses to hepatitis C.

...

DETAILED DESCRIPTION:
S-adenosyl methionine (SAMe) is a nutritional supplement which is available as an over-the-counter formula. It is a naturally occurring, modified amino acid that is produced in virtually all cells and participates in many biochemical pathways as a major methyl donor and may play a role in intracellular interferon signaling.

This study will assess the effects of SAMe on antiviral responses to peginterferon and ribavirin in patients with chronic hepatitis C, genotype 1, who have failed to respond to a previous course of therapy. After screening evaluation, patients will receive a first course of 2 weeks of peginterferon alfa-2a (180 micrograms weekly) and ribavirin (1000-1200 mg daily) during which symptoms, routine laboratory tests, HCV RNA levels, natural killer (NK) cell activity, and lymphocyte interferon-signaling responses will be monitored. After a 4-week washout period, patients will start SAMe (800 mg twice daily) for 2 weeks and then begin a second course of peginterferon and ribavirin in the same doses with similar monitoring. Therapy will be continued for at least 12 weeks, and patients with an early viral response will continue for a full 48 weeks. The primary criterion for efficacy of SAMe will be improved HCV kinetic responses comparing the first and second courses of peginterferon and ribavirin. Secondary endpoints will be improvement in NK cell activity and intracellular interferon signaling.

This is a pilot study to determine whether SAMe improves responses to peginterferon therapy in terms of intracellular interferon signaling, innate immune responses, and decline in viral levels.

ELIGIBILITY:
INCLUSION CRITERIA

* Age 18 years or above, male or female
* Serum alanine or aspartate aminotransferase (ALT & AST) activities that are above the upper limit of normal (ALT greater than 41 or AST greater than 31 IU/L).
* Presence of anti-HCV in serum.
* Presence of HCV RNA genotype 1 in serum at levels above 10,000 copies/ml.
* Previous adequate therapy with interferon and ribavirin or peginterferon and ribavirin without a sustained virological response. An adequate course of therapy is defined as at least 12 weeks of interferon in doses of 3 million units three times weekly or peginterferon in doses of 180 micrograms for peginterferon alfa-2a or 1.5 micrograms/kg for peginterferon alfa 2b once weekly and ribavirin in starting doses of at least 1000 mg daily. Patients who initiated therapy at these doses, but required dose modification due to side effects will also be eligible.
* Written informed consent: Patients will be informed of the risk/benefits and side-effects of the medications used in this protocol and will be advised of the research blood drawn at each clinic visit. They will be given ample time to read the consent form and to ask any protocol related questions. Once this is done, the patient's signature will be obtained on the consent form to enroll them into the protocol.

EXCLUSION CRITERIA

* Evidence of other forms of liver disease.
* Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg) in serum.
* Primary sclerosing cholangitis as defined by liver histology.
* Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
* Autoimmune hepatitis as defined by antinuclear antibody (ANA) of 3 EU or greater (ELISA) and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy for autoimmune hepatitis.
* Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
* Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D. Patients with iron saturation indices of greater than 45% and serum ferritin levels of greater than 300 ng/ml for men and greater than 250 ng/ml for women will undergo genetic testing for C282Y and H63D.
* Drug induced liver disease as defined on the basis of typical exposure and history.
* Bile duct obstruction as suggested by imaging studies done within the previous six months.
* Decompensated liver disease, as marked by bilirubin greater than 4 mg/dl, albumin less than 3.0 gm/l, prothrombin time greater than 2 sec prolonged, Child-Pugh score of 7 or greater or history of bleeding esophageal varices, ascites or hepatic encephalopathy. Patients with ALT levels greater than 1000 U/L (greater than 25 times the upper limit of the normal range) will not be enrolled but may be followed until three determinations are below this level.
* Significant systemic or major illnesses other than liver disease, including congestive heart failure, coronary artery disease, cerebrovascular disease, pulmonary disease with hypoxia, renal failure, organ transplantation, serious psychiatric disease including depression, malignancy and any other conditions that in the opinion of the investigator would preclude treatment.
* Pre existing, severe bone marrow compromise; anemia (hematocrit less than 34%), neutropenia (less than 1000 polymorphonuclear cells/mm(3)) or thrombocytopenia (less than 70,000 cells/mm(3)).
* Serious autoimmune disease that, in the opinion of the investigators, might be worsened by interferon therapy, such as lupus erythematous, rheumatoid arthritis or Crohn's disease
* Known HIV infection.
* Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year.
* Pregnancy, lactation or in women of child bearing potential or in spouses of such women, inability to practice adequate contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicide, birth control pills/depot injection, or an intrauterine device.
* Evidence of hepatocellular carcinoma; either alpha-fetoprotein (AFP) levels greater than 50 ng/ml (normal less than 9 ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.
* Immunosuppressive therapy with either corticosteroids (more than 5 mg of prednisone daily) or major immunosuppressive agents (such as azathioprine or 6-mercaptopurine).
* Clinical gout at presentation.
* History of hypersensitivity reactions to S-adenosyl methionine.
* Serum creatinine greater than 1.5mg/dl in men and greater than 1.4 mg/dl for women.
* Any other condition, which in the opinion of the investigators would impede the patient's participation or compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hoofnagle, MD, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Thomas DL, Seeff LB. Natural history of hepatitis C. Clin Liver Dis. 2005 Aug;9(3):383-98, vi. doi: 10.1016/j.cld.2005.05.003. PMID 16023972
- [Derived] Feld JJ, Modi AA, El-Diwany R, Rotman Y, Thomas E, Ahlenstiel G, Titerence R, Koh C, Cherepanov V, Heller T, Ghany MG, Park Y, Hoofnagle JH, Liang TJ. S-adenosyl methionine improves early viral responses and interferon-stimulated gene induction in hepatitis C nonresponders. Gastroenterology. 2011 Mar;140(3):830-9. doi: 10.1053/j.gastro.2010.09.010. Epub 2010 Sep 17. PMID 20854821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four patients were enrolled at National Institutes of Health Clinic Center between October 2007 and April 2009.
Groups:
- Hepatitis C Treated With Peginterferon and Ribavirin: Patients infected with hepatitis C virus (HCV) treated with peginterferon alpha-2a and ribavirin. After screening evaluation, patients will receive a first course of 2 weeks of peginterferon alfa-2a (180 micrograms weekly) and ribavirin (1000-1200 mg daily) during which symptoms, routine laboratory tests, HCV RNA levels, natural killer (NK) cell activity, and lymphocyte interferon-signaling responses will be monitored. After a 4-week washout period, patients will start SAMe (800 mg twice daily) for 2 weeks and then begin a second course of peginterferon and ribavirin in the same doses with similar monitoring. Therapy will be continued for at least 12 weeks, and patients with an early viral response will continue for a full 48 weeks.
Period: Overall Study
Arm/Group | Hepatitis C Treated With Peginterferon and Ribavirin
Started | 24
Completed | 20
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Hepatitis C Treated With Peginterferon and Ribavirin: Patients infected with hepatitis C virus (HCV) treated with peginterferon alpha-2a and ribavirin
Arm/Group | Hepatitis C Treated With Peginterferon and Ribavirin
Number analyzed (Participants) | 24
Age Continuous [Median (Full Range); unit: year] | 52.5 [41 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race/Ethnicity, Customized [Number; unit: participants] — Race
  participants
    Hispanic | 1
    Black | 2
    White | 21
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (3.74)
Ishak Fibrosis [Median (Full Range); unit: Units on a scale] — Possible range is 0 to 6. Higher values represent worse outcomes.
  Units on a scale | 2 [0 to 6]
Cirrhosis [Number; unit: participants]
  Cirrhosis | 5
  Non-Cirrhosis | 19
Previous Therapy [Number; unit: participants]
  Interferon/ribavirin | 3
  Peginterferon/ribavirin | 21
Baseline HCV RNA Level [Mean (Standard Deviation); unit: log10 (IU/mL)] | 6.3 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Viral Kinetics During the First 2 Weeks of Therapy
Description: Improvement of slopes of decline in hepatitis C virus Ribonucleic acid in second course compared with first course in days 7 to 14 of therapy
Time Frame: Days 7 to 14 of therapy
Population: Of 24 patients enrolled, 3 patients completed first course only due to adverse effects or personal reason. A fourth patient completed both courses but missed blood draws in both courses, precluding calculation of accurate first- and second-phase kinetic parameters. These 4 patient were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Hepatitis C Treated With Peginterferon and Ribavirin
Number analyzed (Participants) | 20
participants | 14

2. Secondary Outcome: 2-log Decline in HCV RNA by Week 12 (Early Virological Response) and Sustained Eradication of HCV RNA (Sustained Virological Response).
Description: 2-log decline in HCV RNA by week 12 (early virological response) and sustained eradication of HCV RNA (sustained virological response).
Time Frame: 12 weeks from start of therapy
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Hepatitis C Treated With Peginterferon and Ribavirin
Number analyzed (Participants) | 20
participants | 11

ADVERSE EVENTS:
Arm/Group | Hepatitis C Treated With Peginterferon and Ribavirin
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatitis C Treated With Peginterferon and Ribavirin (N=24)
Rash attributed to ribavirin (Skin and subcutaneous tissue disorders) | 1 (1)
Benzodiazepine abuse (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes